CLINICAL TRIAL: NCT02822040
Title: An Evaluation of Root Length Measurements Using Intraoral Scan and Panoramic
Brief Title: An Evaluation of Root Length Measurements Using Intraoral Scan and Panoramic Radiographs
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Rodrigo Viecilli, DDS, PhD, Orthodontic Faculty, Loma Linda University
Other Study IDs: 5160149
Record Dates: First submitted 2016-04-18; First posted 2016-07-04 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Root Resorption
Keywords: Root Resorption; Panoramic Radiograph
MeSH Terms: conditions — Root Resorption

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Experimental group: All patients who have initial and final records qualify in the experimental group.
  Interventions: Other: Intraoral Scan

INTERVENTIONS:
Other: Intraoral Scan — All patients will have an intraoral scan performed for measurements to be taken on.

SUMMARY:
This study will attempt to validate a method of estimating root length on panoramic radiograph by crown measurement on intraoral digital scans.

DETAILED DESCRIPTION:
Intraoral digital scans will be taken on patients who have completed orthodontic treatment, and measurements will be made on the crown dimensions. These dimensions will then be applied onto the same teeth as seen on panoramic radiographs and a mathematical relationship will be determined for root length. Changes in root length will be measured from initial records to treatment complete panoramic radiographs and these estimates will be compared to actual root length changes as measured in CBCT (Cone Beam Computed Tomography) records.

ELIGIBILITY:
Inclusion Criteria:

* Subject has initial records including CBCT scan and panoramic radiograph that are clear. Subject must have no restorations or significant loss in tooth structure in target teeth or teeth adjacent to target.

Exclusion Criteria:

* Subjects who have records that are not clear, and who are missing target teeth.

Ages: 13 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who have undergone orthodontic treatment, and associated tooth movement, and have initial records directly before the initiation of treatment.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in root length in mm | Root length will be measured at the initiation of orthodontic treatment and at an average of 24 months later.
  Changes in root length will be calculated, starting from the initiation of orthodontic treatment to completion of treatment, at an average of 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Viecilli, DDS, PhD, Principal Investigator — Loma Linda University

IPD SHARING:
Plan to Share IPD: No